CLINICAL TRIAL: NCT07357181
Title: Impact of Manual Preference on Motor Deficits After Stroke
Brief Title: Influence of Handedness on Upper Limb Recovery
Acronym: HANDISTROKE
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Other Study IDs: CHUO-2025-19
Record Dates: First submitted 2026-01-13; First posted 2026-01-21 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Stroke
Keywords: Stroke; Handedness; Motricity; Upper Limb; Manual preference; Motor impairment; Motor recovery
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with confirmed unilateral recent stroke
  Interventions: Other: evaluation

INTERVENTIONS:
Other: evaluation — Patients will be evaluated at baseline for Edinburgh Handedness Inventory Laterality Quotient. Patients will be seen again at 6 months as part of their standard post-stroke consultation at Orléans University Hospital by a neurologist from the neurology department. In conjunction with this consultation, an assessment specific to this research study of the FMA-UE and SAFE scores will be carried out by a physiotherapist from the department.

SUMMARY:
This prospective, single-center observational study evaluates whether handedness is associated with upper-limb motor recovery after a recent unilateral stroke. Adults admitted to the stroke unit with a confirmed unilateral stroke within 5 days are included if they do not object to participation. Upper-limb impairment is assessed early after stroke and at 6 months using standardized clinical scales. Handedness is determined by self-report, and the Edinburgh Handedness Inventory is administered when feasible. The main hypothesis is that left-handed participants may show better upper-limb motor recovery at 6 months than right-handed participants, potentially due to differences in brain motor network lateralization.

DETAILED DESCRIPTION:
Participants hospitalized in the stroke unit with a confirmed unilateral stroke are recruited consecutively. After eligibility verification and absence of objection, baseline data are collected within 5 days post-stroke. Baseline assessments include the Fugl-Meyer Assessment for the Upper Extremity (FMA-UE), the Shoulder Abduction and Finger Extension (SAFE) score, and the National Institutes of Health Stroke Scale (NIHSS) score (post-acute treatment if thrombolysis or thrombectomy was performed). Handedness is recorded after the motor assessments to maintain assessor blinding regarding group membership; the Edinburgh Handedness Inventory is administered when cognitive status allows. A 6-month follow-up is performed during routine post-stroke consultation at the study site, with repeat FMA-UE and SAFE assessments. The primary analysis compares FMA-UE at 6 months between left-handed and right-handed participants among those with baseline FMA-UE less than 66, using propensity score matching (3:1 right-handed to left-handed) accounting for age, baseline motor deficit, lesion side relative to dominance (dominant vs non-dominant hemisphere), and stroke type (ischemic vs hemorrhagic).

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed unilateral recent stroke (less than 5 days).
2. Age 18 years and older.
3. Participant or proxy does not object to participation

Exclusion Criteria:

1. Prior stroke with residual motor sequelae.
2. Pre-stroke upper-limb deficit.
3. Follow-up at 6 months not planned at Orléans.
4. Protected adult (guardianship/curatorship), person under legal protection, or deprived of liberty.
5. Pregnant or breastfeeding woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults hospitalized in the stroke unit of Orléans University Hospital with a confirmed unilateral recent stroke.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment for Upper Extremity (FMA-UE) Score | month 6
  Upper-limb motor impairment measured using the Fugl-Meyer Assessment for the Upper Extremity (FMA-UE) at 6 months post-stroke. Scores range from 0 to 66, with higher scores indicating less impairment. Primary analysis is performed among participants with baseline FMA-UE less than 66.

SECONDARY OUTCOMES:
Mean Fugl-Meyer Assessment for Upper Extremity (FMA-UE) Score | Baseline
  Score from 0 to 66; the lower the score, the more severe the deficit
Proportion of Left-Handed Participants | Baseline
Mean National Institutes of Health Stroke Scale (NIHSS) Score | Baseline
  Score from 0 to 42; the higher the score, the more severe the deficit
Number of Participants With Upper-Limb Weakness | Baseline
  Number of Participants With Upper-Limb Weakness Defined as SAFE Score Less Than 10
Correlation Between Edinburgh Handedness Inventory Laterality Quotient and Baseline FMA-UE Score | Baseline
  Score from -100 to +100, no notion of severity here since it assesses manual preference (at -100 you are very left-handed and at +100 you are very right-handed)
Mean Shoulder Abduction and Finger Extension (SAFE) Score | Month 6
  Score from 0 to 10; the lower the score, the more severe the deficit.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Orléans, Orléans, France

REFERENCES:
- [Background] Harris JE, Eng JJ. Individuals with the dominant hand affected following stroke demonstrate less impairment than those with the nondominant hand affected. Neurorehabil Neural Repair. 2006 Sep;20(3):380-9. doi: 10.1177/1545968305284528. PMID 16885424
- [Background] Papadatou-Pastou M, Ntolka E, Schmitz J, Martin M, Munafo MR, Ocklenburg S, Paracchini S. Human handedness: A meta-analysis. Psychol Bull. 2020 Jun;146(6):481-524. doi: 10.1037/bul0000229. Epub 2020 Apr 2. PMID 32237881
- [Background] Bonnal J, Pila O, Papin C, Lebkowski L, Sarrazin M, Bravo R, Prieur F. Handedness and task demands modulate motor cortex lateralization: A cross-sectional fNIRS study. Neuroimage. 2025 Dec 1;323:121578. doi: 10.1016/j.neuroimage.2025.121578. Epub 2025 Nov 9. PMID 41218702
- [Background] Tzourio-Mazoyer N, Petit L, Zago L, Crivello F, Vinuesa N, Joliot M, Jobard G, Mellet E, Mazoyer B. Between-hand difference in ipsilateral deactivation is associated with hand lateralization: fMRI mapping of 284 volunteers balanced for handedness. Front Hum Neurosci. 2015 Feb 6;9:5. doi: 10.3389/fnhum.2015.00005. eCollection 2015. PMID 25705184
- [Background] Darling WG, Helle N, Pizzimenti MA, Rotella DL, Hynes SM, Ge J, Stilwell-Morecraft KS, Morecraft RJ. Laterality affects spontaneous recovery of contralateral hand motor function following motor cortex injury in rhesus monkeys. Exp Brain Res. 2013 Jul;228(1):9-24. doi: 10.1007/s00221-013-3533-1. Epub 2013 May 8. PMID 23652723
- [Background] Solodkin A, Hlustik P, Noll DC, Small SL. Lateralization of motor circuits and handedness during finger movements. Eur J Neurol. 2001 Sep;8(5):425-34. doi: 10.1046/j.1468-1331.2001.00242.x. PMID 11554905